CLINICAL TRIAL: NCT01459601
Title: Cabergoline Effects on Blood Sugar Control in Type 2 Diabetics
Brief Title: Cabergoline Effect on Blood Sugar in Type 2 Diabetics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Haleh Rokni Yazdi, assisstant professor, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CabergolinDM
Record Dates: First submitted 2011-10-24; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Diabetes Type 2
Keywords: diabetes mellitus; FBS; HbA1C; Cabergoline
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Cabergoline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cabergoline — 0,5mg per week
  Other Names: Dastinex

SUMMARY:
Diabetic patients with poorly control blood sugar are prescribed cabergoline for 1 months and their blood glucose is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1C>7

Exclusion Criteria:

* HbA1C>10
* Psychiatric disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
FBS (fasting blood sugar) | 30days

SECONDARY OUTCOMES:
HbA1C | 30days